CLINICAL TRIAL: NCT03548402
Title: Acceptance and Commitment Therapy for Nonsuicidal Self-injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Heather McClary, Director of Research Compliance, Southern Methodist University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-029-MEUA
Record Dates: First submitted 2013-05-10; First posted 2018-06-07 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Nonsuicidal Self-Injury; Anxiety
MeSH Terms: conditions — Self-Injurious Behavior; Anxiety Disorders | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT is based on the theory that rigid attempts to control internal states, thoughts and feelings, and other forms of experiential avoidance contribute to symptom development and maintenance of anxiety and self-injury.

SUMMARY:
The goal of this study is to evaluate the effectiveness of Acceptance and Commitment Therapy (ACT) for individuals who engage in nonsuicidal self-injury(NSSI) and have comorbid anxiety.

With the data collected from the study, the investigators will test the following hypotheses:

Acceptance and commitment therapy will lead to reductions in anxiety and self-harm behaviors in non-suicidal self-injury individuals.

DETAILED DESCRIPTION:
Non-suicidal self-injury is the direct and purposeful harming of one's bodily tissue outside of social and religious norms and lacking suicidal intent. The most common NSSI behaviors include cutting (70-90%), banging or hitting (21-44%), and burning (15-35%) (Rodham & Hawton, 2009); but many report utilizing multiple methods (50-70%; Klonsky, 2011; Whitlock, Eckenrode, & Silverman, 2006). NSSI has an alarming prevalence among college students, with rates ranging from 17-38% (Whitlock et al., 2006; Gratz, Conrad, & Roemer, 2002). NSSI occurs in the context of many psychological disorders (Nock, 2010), and is associated with anxiety and mood disturbances (Andover et al., 2005). This is a prevalent problem and lacks an efficacious treatment. As a result, this study can shed insight into possible treatments.

The experiential avoidance model of deliberate self-harm posits that a function of self-injury is maintained through negative reinforcement by reducing unpleasant emotional arousal (Chapman et al. 2006). Therefore a treatment that directly targets reducing experiential avoidance is likely to be effective.

ACT is based on the theory that rigid attempts to control internal states, thoughts and feelings, and other forms of experiential avoidance contribute to symptom development and maintenance of anxiety and self-injury. The training includes three components: (a) educating Ps about the exacerbation of anxiety symptoms and problem behaviors through rigid attempts at experiential avoidance, (b) introducing acceptance and the willingness to experience anxiety-related sensations and cognitions as an alternative to experiential control, through the practice of intentional and non-judgmental paying attention to one's thoughts, feelings, images and bodily sensations (including aversive symptoms of anxiety) and learning to see thoughts as an ongoing process distinct from self rather than merely an event with literal meaning (cognitive defusing), and (c) instructing Ps in between-session exercises incorporating awareness of present, internal experiences and cognitive defusion exercises while engaging in exercises that give rise to them.

ELIGIBILITY:
Inclusion Criteria:

1. If applicable, be stabilized on their current medications for at least two months.
2. Must report at least one incidence of self-injuring during the past six months.

Exclusion Criteria:

* Active psychosis, schizophrenia and schizoaffective disorder Current active suicidal ideation Individuals with a history of seizure disorders, angina, myocardial infarction, congestive heart failure, clinically significant arrhythmias, transient ischemic attacks, cerebrovascular accidents, diabetes mellitus, significant asthma, emphysema, chronic obstructive pulmonary disease or a family history of heart disease before age 55 are also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03-19 (Actual); Primary Completion 2015-03-19 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Urges to Self-Injure | During treatment (weeks 1-10) and 2 month follow-up
  Whether there is a decrease in the participants self-reported urge to self-injure as measured by the Alexian Brothers Urge to Self-Injure Scale (ABUSI). Responses are on a 7-point scale with a maximum total score of 30 and higher scores reflecting more intense urges to self-injure.

SECONDARY OUTCOMES:
Experiential Avoidance | During treatment (weeks 1-10) and at 2 month follow-up
  Whether there are reductions in the participants self-reported experiential avoidance measured by the Acceptance and Action Questionnaire-II (AAQ-II)

OTHER OUTCOMES:
Anxiety | During treatment (weeks 1-10) and at 2 month follow-up
  Whether there are changes in the participants self-reported anxiety symptoms measured by the Anxiety Sensitivity Index (ASI)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Meuret, PhD, Principal Investigator — Southern Methodist University
Locations (1):
- Stress, Anxiety, and Chronic Disease Research Program, Southern Methodist University, Dallas, Texas, United States

REFERENCES:
- [Background] Washburn JJ, Juzwin KR, Styer DM, Aldridge D. Measuring the urge to self-injure: preliminary data from a clinical sample. Psychiatry Res. 2010 Aug 15;178(3):540-4. doi: 10.1016/j.psychres.2010.05.018. Epub 2010 Jun 30. PMID 20580437